CLINICAL TRIAL: NCT06891040
Title: A Multicenter, Randomized, Double-blind, Vehicle Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of VC005 in Adult Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of VC005 in Adult Subjects With Mild to Moderate Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-203
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VC005 Low Dose groups (Experimental): VC005 group with Local topical application
  Interventions: Drug: VC005 groups
- VC005 high Dose groups (Experimental): VC005 group with Local topical application
  Interventions: Drug: VC005 groups
- VC005 Placebo groups (Placebo Comparator): VC005 Placebo group with Local topical application
  Interventions: Drug: VC005 Placebo group

INTERVENTIONS:
Drug: VC005 Placebo group — VC005 Placebo group with Local topical application
  Arms: VC005 Placebo groups
Drug: VC005 groups — VC005 group with Local topical application
  Arms: VC005 Low Dose groups; VC005 high Dose groups

SUMMARY:
A multicenter, randomized, double-blind, vehicle controlled phase II clinical study

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand this study, are able to follow the relevant procedures of the trial, voluntarily participate in the clinical trial, and sign the informed consent form (ICF);
2. The age requirement for signing the ICF is 18 years old or above, with no gender restrictions;
3. During screening, the diagnosis of atopic dermatitis should be met according to the Hanifin-Rajka criteria;

Exclusion Criteria:

1. Skin damage or abnormalities that may affect the evaluation of the administration site of the investigational drug;
2. Skin diseases that are contraindicated in research or affect the evaluation of drug administration sites, including but not limited to psoriasis, acne, and skin cancer;
3. Suffering from autoimmune diseases other than AD, such as inflammatory bowel disease and rheumatoid arthritis, and the researchers believe that this disease will be detrimental to the evaluation of this study;
4. Current history of or presence of lymphoproliferative disorders, or signs or symptoms suggesting possible lymphoproliferative disorders, including lymphadenopathy or splenomegaly;
5. Various malignant tumors, or any history of malignant tumors within the past 5 years prior to screening (excluding completely resected cervical carcinoma in situ, non metastatic squamous cell carcinoma, basal cell carcinoma, or papillary thyroid carcinoma);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in EASI（Eczema area and severity index） from baseline | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Qian jin Lu, Principal Investigator — Chinese Academy of Medical Sciences Hospital of Skin Disease
Locations (1):
- Chinese Academy of Medical Sciences Hospital of Skin Disease, Nanjing, Jiangsu, China